CLINICAL TRIAL: NCT00509769
Title: A Phase II, Single-arm, Open-label Study of Trastuzumab-MCC-DM1 Administered Intravenously to Patients With HER2-Positive Metastatic Breast Cancer Who Have Progressed While Receiving HER2-Directed Therapy
Brief Title: A Study of Trastuzumab Emtansine (Trastuzumab-MCC-DM1) Administered Intravenously to Patients With Human Epidermal Growth Factor Receptor 2 (HER2)-Positive Metastatic Breast Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TDM4258g
Record Dates: First submitted 2007-07-27; First posted 2007-07-31 (Estimated); Results first posted 2013-04-02 (Estimated); Last update posted 2013-04-02 (Estimated); Status verified 2013-02

CONDITIONS: Metastatic Breast Cancer
Keywords: Trastuzumab emtansine; MBC; Breast cancer; HER2-positive breast cancer; HER2
MeSH Terms: conditions — Breast Neoplasms | interventions — Ado-Trastuzumab Emtansine

ARMS (1):
- Trastuzumab emtansine 3.6 mg/kg (Experimental): Patients received trastuzumab emtansine 3.6 mg/kg intravenously on Day 1 of each 21 day cycle for a maximum of 1 year. The total dose was dependent on the patient's weight on Day 1 of each cycle.
  Interventions: Drug: Trastuzumab emtansine [Kadcyla]

INTERVENTIONS:
Drug: Trastuzumab emtansine [Kadcyla] — Trastuzumab emtansine was provided in either a liquid or a lyophilized formulation.
  Other Names: trastuzumab-DM1; trastuzumab-MCC-DM1; T-DM1

SUMMARY:
This was a multi-institutional, open-label, single-arm, Phase II study of trastuzumab emtansine (T-DM1) administered by intravenous (IV) infusion to patients with human epidermal growth factor receptor 2 (HER2)-positive metastatic breast cancer (MBC).

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent form.
* Human epidermal growth factor receptor 2 (HER2)-positive metastatic breast cancer (MBC); tissue (slides or blocks) available for HER2 confirmation.
* History of progression on HER2-directed therapy for the treatment of HER2-positive breast cancer.
* At least 1, and no more than 3, chemotherapy regimens for MBC.
* Granulocyte count ≥ 1500/μL, platelet count ≥ 100,000/μL, and hemoglobin ≥ 9 g/dL.
* Serum bilirubin ≤ 1.5 mg/dL, aspartate aminotransferase (AST), alanine aminotransferase (ALT), and alkaline phosphatase ≤ 2.5x the upper limit of normal (ULN).
* Serum creatinine ≤ 1.5 mg/dL or creatinine clearance ≥ 60 mL/min.
* Eastern Cooperative Oncology Group (ECOG) performance status of 0, 1, or 2.

Exclusion Criteria:

* Any chemotherapy, hormonal therapy, radiotherapy, immunotherapy, or biological therapy for the treatment of breast cancer within 2 weeks of the first study treatment.
* Prior cumulative doxorubicin dose > 360 mg/m^2 or the equivalent.
* History of significant cardiac disease, unstable angina, congestive heart failure (CHF), myocardial infarction, or ventricular arrythmia requiring medication.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 112 (Actual)
Dates: Start 2007-07; Primary Completion 2009-01 (Actual); Study Completion 2009-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Scott Holden, M.D., Study Director — Genentech, Inc.
Locations (40):
- United States (40):
  - Little Rock Hem Onc Assoc, Little Rock, Arkansas
  - Rocky Mountain Cancer Center, Denver, Colorado
  - Washington Cancer Institute, Washington D.C., District of Columbia
  - Lynn Cancer Institute - West, Boca Raton, Florida
  - Florida Cancer Care, Davie, Florida
  - Mayo Clinic, Jacksonville, Florida
  - Hem/Onc Assoc - Treasure Coast, Port Saint Lucie, Florida
  - Gulfcoast Oncology Associates, St. Petersburg, Florida
  - Bay Area Oncology, Tampa, Florida
  - Northwest Georgia Onc Ctrs PC, Marietta, Georgia
  - John McClean, M.D. - Private P, Galesburg, Illinois
  - Cedar Valley Med Specialists, Waterloo, Iowa
  - Kentuckiana Cancer Institute, Louisville, Kentucky
  - Minnesota Oncology Hematology,, Minneapolis, Minnesota
  - Missouri Cancer Associates, Columbia, Missouri
  - Kansas City Cancer Center, LLC, Lee's Summit, Missouri
  - St. Louis Cancer & Breast Inst, St Louis, Missouri
  - St. Barnabas Health Care Sys, Livingston, New Jersey
  - New York Oncology Hematology, Albany, New York
  - Eastchester Center/Cancer Care, The Bronx, New York
  - Carolinas Hem-Oncology Assoc, Charlotte, North Carolina
  - Raleigh Hemotology & Oncology, Raleigh, North Carolina
  - Midwestern Regional Med Center, Eugene, Oregon
  - Texas Oncology Cancer Center, Austin, Texas
  - Texas Oncology, P.A., Bedford, Texas
  - Cancer Specialists of South Te, Corpus Christi, Texas
  - US Oncology Research, Inc., Dallas, Texas
  - USO, Dallas, Texas
  - Texas Oncology, P.A., Dallas, Texas
  - Sammons Cancer Center, Dallas, Texas
  - El Paso Cancer Treatment Ctr, El Paso, Texas
  - Texas Oncology PA, Fort Worth, Texas
  - Texas Oncology, P.A., Houston, Texas
  - US Oncology, Midland, Texas
  - USO - Tyler Cancer Ctr, Tyler, Texas
  - Waco Cancer Care & Research Ce, Waco, Texas
  - Northern Utah Associates, Ogden, Utah
  - Fairfax N Virginia Hem/Onc PC, Fairfax, Virginia
  - Northwest Medical Specialties, Tacoma, Washington
  - Northwest Cancer Specialists, Vancouver, Washington

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Trastuzumab Emtansine 3.6 mg/kg
Started | 112
Completed | 21
Not Completed | 91
Not completed — Progressive disease | 77
Not completed — Adverse Event | 4
Not completed — Patient's decision | 1
Not completed — Physician Decision | 8
Not completed — Use of prohibited therapies during study | 1

BASELINE CHARACTERISTICS:
Arm/Group | Trastuzumab Emtansine 3.6 mg/kg
Number analyzed (Participants) | 112
Age Continuous [Mean (Standard Deviation); unit: years] | 55.0 (10.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 111
  Male | 1

OUTCOME MEASURES:

1. Primary Outcome: Objective Response Assessed by the Independent Review Facility Using Response Evaluation Criteria in Solid Tumors (RECIST)
Description: Objective response was defined as a complete response (CR) or partial response (PR) determined on 2 consecutive occasions ≥ 4 weeks apart, using Response Evaluation Criteria in Solid Tumors (RECIST). CR: The disappearance of all target lesions and all non-target lesions, normalization of tumor marker level, and no new lesions. PR: Disappearance of all target lesions and persistence of ≥ 1 non-target lesions and/or the maintenance of tumor marker level above the normal limits, or, at least a 30% decrease in the sum of the longest diameter of target lesions, and no new lesions or unequivocal progression of existing non-target lesions.
Time Frame: Randomization until the analysis data cutoff-dates of 31 Jan 2009 (6 months after the last patient was enrolled in the study) and 25 Jun 2009 (approximately 12 months after the last patient was enrolled in the study, up to 23 months)
Population: Efficacy evaluable population: All patients who received at least 1 dose of study drug and who underwent a baseline and at least 1 post-baseline tumor assessment or died while in the study from any cause within 30 days of the last dose of study drug.
Measure: Number (95% Confidence Interval); unit: Percentage of patients
Arm/Group | Trastuzumab Emtansine 3.6 mg/kg
Number analyzed (Participants) | 109
Percentage of patients
  Month 6 (n=109) | 25.7 [17.9 to 34.5]
  Month 12 (n=108) | 26.9 [19.2 to 35.8]

2. Secondary Outcome: Duration of Objective Response (OR) Assessed by the Independent Review Facility Using Response Evaluation Criteria in Solid Tumors (RECIST)
Description: For patients who achieved an objective response, duration of objective response was defined as the time from the first tumor assessment that supported a patient's objective response to the time of disease progression or death on study (ie, death from any cause within 30 days of the last dose of study drug), whichever occurred first. Disease progression was defined as at least a 20% increase in the sum of the longest diameter of target lesions, taking as reference the smallest sum longest diameter recorded since treatment started or the appearance of 1 or more new lesions or the appearance of 1 or more new lesions and/or unequivocal progression of existing non-target lesions. For participants who experienced no disease progression and did not die while on study, data were censored at the date of the last tumor assessment. Kaplan-Meier methodology was used to estimate the duration of objective response.
Time Frame: Randomization until the final analysis cut-off date of 25 Jun 2009 (end of the study, approximately 12 months after the last patient was enrolled, up to 23 months)
Population: Patients who had an objective response in the efficacy evaluable population: All patients who received at least 1 dose of study drug and who underwent a baseline and at least 1 post-baseline tumor assessment or died while in the study from any cause within 30 days of the last dose of study drug.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Trastuzumab Emtansine 3.6 mg/kg
Number analyzed (Participants) | 108
Months | NA [6.2 to NA] — The median and the upper limit of the 95% confidence interval were not reached because of insufficient events.

3. Secondary Outcome: Progression-free Survival (PFS) Assessed by the Independent Review Facility Using Response Evaluation Criteria in Solid Tumors (RECIST)
Description: Progression-free survival (PFS) was defined as the time from the first day of study treatment to documented disease progression or death on study (ie, death from any cause within 30 days of the last dose of study drug), whichever occurred first. Disease progression was at least a 20% increase in the sum of the longest diameter of target lesions, taking as reference the smallest sum longest diameter recorded since the treatment started or the appearance of 1 or more new lesions or the appearance of 1 or more new lesions and/or unequivocal progression of existing non-target lesions. For patients who experienced no disease progression and did not die while on study, data were censored at the date of the last tumor assessment. Kaplan-Meier methodology was used to estimate PFS.
Time Frame: as for outcome 2
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Trastuzumab Emtansine 3.6 mg/kg
Number analyzed (Participants) | 108
Months | 4.6 [3.9 to 8.6]

4. Secondary Outcome: Objective Response Determined by the Investigator Using Response Evaluation Criteria in Solid Tumors (RECIST)
Description: as for outcome 1
Time Frame: as for outcome 2
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of patients
Arm/Group | Trastuzumab Emtansine 3.6 mg/kg
Number analyzed (Participants) | 108
Percentage of patients | 38.9 [29.7 to 48.5]

5. Secondary Outcome: Duration of Objective Response Assessed by the Investigator Using Response Evaluation Criteria in Solid Tumors (RECIST)
Description: as for outcome 2
Time Frame: as for outcome 2
Population: as for outcome 2
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Trastuzumab Emtansine 3.6 mg/kg
Number analyzed (Participants) | 108
Months | 9.4 [7.0 to NA] — The upper limit of the 95% confidence interval were not reached because of insufficient events.

6. Secondary Outcome: Progression-free Survival Assessed by the Investigator Using Response Evaluation Criteria in Solid Tumors (RECIST)
Description: as for outcome 3
Time Frame: as for outcome 2
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Trastuzumab Emtansine 3.6 mg/kg
Number analyzed (Participants) | 108
Months | 4.6 [4.1 to 6.0]

ADVERSE EVENTS:
Time Frame: Adverse events were recorded from randomization through the end of the study.
Description: Safety population: All patients who received any amount of trastuzumab emtansine.
Arm/Group | Trastuzumab Emtansine 3.6 mg/kg
Serious Adverse Events (participants affected / at risk) | 30/112
Other Adverse Events (participants affected / at risk) | 110/112
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Trastuzumab Emtansine 3.6 mg/kg (N=112)
Thrombocytopenia (Blood and lymphatic system disorders) | 1
Dysphagia (Gastrointestinal disorders) | 1
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 1
Oesophageal stenosis (Gastrointestinal disorders) | 1
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1
Asthenia (General disorders) | 1
Disease progression (General disorders) | 1
Hepatotoxicity (Hepatobiliary disorders) | 1
Cellulitis (Infections and infestations) | 3
Pneumonia (Infections and infestations) | 2
Osteomyelitis (Infections and infestations) | 1
Urosepsis (Infections and infestations) | 1
Hip fracture (Injury, poisoning and procedural complications) | 1
Subdural haemorrhage (Injury, poisoning and procedural complications) | 1
Hepatic enzyme increased (Investigations) | 1
Platelet count decreased (Investigations) | 1
White blood cell count increased (Investigations) | 1
Dehydration (Metabolism and nutrition disorders) | 1
Failure to thrive (Metabolism and nutrition disorders) | 1
Back pain (Musculoskeletal and connective tissue disorders) | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 1
Groin pain (Musculoskeletal and connective tissue disorders) | 1
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1
Acute myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Convulsion (Nervous system disorders) | 2
Altered state of consciousness (Nervous system disorders) | 1
Aphasia (Nervous system disorders) | 1
Cerebrovascular accident (Nervous system disorders) | 1
Confusional state (Psychiatric disorders) | 2
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1
Deep vein thrombosis (Vascular disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Trastuzumab Emtansine 3.6 mg/kg (N=112)
Anaemia (Blood and lymphatic system disorders) | 23
Thrombocytopenia (Blood and lymphatic system disorders) | 18
Neutropenia (Blood and lymphatic system disorders) | 7
Dry eye (Eye disorders) | 11
Lacrimation increased (Eye disorders) | 9
Vision blurred (Eye disorders) | 6
Visual impairment (Eye disorders) | 6
Nausea (Gastrointestinal disorders) | 57
Constipation (Gastrointestinal disorders) | 34
Diarrhoea (Gastrointestinal disorders) | 29
Vomiting (Gastrointestinal disorders) | 27
Dry mouth (Gastrointestinal disorders) | 16
Abdominal pain (Gastrointestinal disorders) | 12
Dyspepsia (Gastrointestinal disorders) | 12
Abdominal pain upper (Gastrointestinal disorders) | 9
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 8
Abdominal discomfort (Gastrointestinal disorders) | 6
Fatigue (General disorders) | 73
Pyrexia (General disorders) | 39
Chills (General disorders) | 22
Pain (General disorders) | 13
Oedema peripheral (General disorders) | 12
Chest pain (General disorders) | 10
Asthenia (General disorders) | 7
Influenza like illness (General disorders) | 7
Infusion related reaction (General disorders) | 7
Upper respiratory tract infection (Infections and infestations) | 20
Urinary tract infection (Infections and infestations) | 18
Contusion (Injury, poisoning and procedural complications) | 12
Weight decreased (Investigations) | 13
Hypokalaemia (Metabolism and nutrition disorders) | 27
Anorexia (Metabolism and nutrition disorders) | 22
Decreased appetite (Metabolism and nutrition disorders) | 16
Dehydration (Metabolism and nutrition disorders) | 6
Pain in extremity (Musculoskeletal and connective tissue disorders) | 25
Arthralgia (Musculoskeletal and connective tissue disorders) | 24
Back pain (Musculoskeletal and connective tissue disorders) | 14
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 13
Myalgia (Musculoskeletal and connective tissue disorders) | 11
Muscle spasms (Musculoskeletal and connective tissue disorders) | 10
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 9
Neck pain (Musculoskeletal and connective tissue disorders) | 8
Muscular weakness (Musculoskeletal and connective tissue disorders) | 6
Headache (Nervous system disorders) | 45
Neuropathy peripheral (Nervous system disorders) | 20
Dizziness (Nervous system disorders) | 13
Dysgeusia (Nervous system disorders) | 7
Insomnia (Psychiatric disorders) | 15
Depression (Psychiatric disorders) | 14
Anxiety (Psychiatric disorders) | 12
Confusional state (Psychiatric disorders) | 7
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 40
Cough (Respiratory, thoracic and mediastinal disorders) | 31
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 23
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 9
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 8
Rash (Skin and subcutaneous tissue disorders) | 19
Pruritus (Skin and subcutaneous tissue disorders) | 8
Hypertension (Vascular disorders) | 7
Hot flush (Vascular disorders) | 6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.